CLINICAL TRIAL: NCT00693875
Title: The Incidence of Intra-Operative Awareness in China and Analysis of Relevant Factors: a Multicentre Study
Status: Completed | Type: Observational
Sponsor: Capital Medical University (Other)
Collaborators: Beijing Chao Yang Hospital (Other); Peking University First Hospital (Other); Peking University Third Hospital (Other); Beijing Friendship Hospital (Other); Beijing Tongren Hospital (Other); Xuanwu Hospital, Beijing (Other); Beijing Hospital (Other Government); China-Japan Friendship Hospital (Other); Beijing Command General Hospital (Unknown); Beijing Obstetrics and Gynecology Hospital (Other); Beijing Hangtian General Hospital (Unknown); Shanghai Rui Jin Hospital (Unknown); Shanghai Zhongshan Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Guangzhou First People's Hospital (Other); Nanfang Hospital, Southern Medical University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); Xijing Hospital (Other); Tang-Du Hospital (Other); Xiangya Hospital of Central South University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Ningbo Medical Center Lihuili Hospital (Other Government); First Hospital of China Medical University (Other); The First Hospital of Jilin University (Other); Fuzhou General Hospital (Other)
Responsible Party: Xu, Liang, BEIJING CHAOYANG HOSPITAL, CAPITAL MEDICAL UNIVERSITY
Other Study IDs: CHAOYANG HOSPITAL
Record Dates: First submitted 2008-06-05; First posted 2008-06-09 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2009-01

CONDITIONS: Intra-Operative Awareness
Keywords: incidence; awareness; general anesthesia; relevant factor; the incidence of intra-operative awareness in China; the relevant factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Medical literature about awareness during general anesthesia is rare in China, and some small sampled studies in China showed a significantly higher incidence (1.5～6%) of intra-operative awareness compared with western countries. The investigators sponsored this multicenter, large sampled, prospective study to determine the incidence of intra-operative awareness in China, and the preservation effect of BIS monitor on the incidence of awareness.

DETAILED DESCRIPTION:
Background: The incidence of awareness in patients undergoing general anesthesia has been reported in as many as 0.1～0.2% in western countries. But so far，medical literature about awareness during general anesthesia is still rare in China, and some small sampled studies in China showed a significantly higher incidence (1.5～6%) of intra-operative awareness. We believed that this multicenter, large sampled, prospective study would be very necessary for us to determine the incidence of intra-operative awareness in China, and analysis of the relevant factors would help us to understand why was the incidence of awareness in China much higher than that in western countries.

Methods: This is a prospective, nonrandomized descriptive cohort study that was conducted at 25 academic medical centers in China. 11,197 patients (age>12, intubation or LMA during anesthesia) form 25 medical centers were enrolled to be interviewed by research stuff for evaluation of awareness at the 1st and 4th day after their general anesthesia. The structured interview questions were:⑴What is the last thing you remembered before you went to sleep? ⑵What is the first thing you remembered when you woke up? ⑶Can you remember anything between these two periods? ⑷Did you dream during your operation? ⑸What was the worst thing about your operation? An evaluation committee independent from the research stuff was constituted to verify the data from the medical centers. And then the incidence of intra-operative awareness in China was determined. General condition and details of the anesthesia procedure of the patients were also recorded during the anesthesia for a binary logistic regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients received general anesthesia with tracheal intubation or LMA
* Apparently normal mental status

Exclusion Criteria:

* Pediatric patients (<12 yr)
* Those who could not be interviewed in 24 hours after the operations
* Those unable to communicate in common spoken Chinese

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subjects would be selected from the patients of the 24 hospitals who would undergo general anesthesia during different kinds of operations in different areas around China after the written informed consents obtained. Each hospital would continuously provide 500～600 subjects for the investigation.
Sampling Method: Probability Sample
Enrollment: 11197 (Actual)
Dates: Start 2007-04; Primary Completion 2008-04 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
evaluation of intra-operative awareness in all the patients investigated | within 4 days after the general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Liang Xu, M.D., Principal Investigator — Capital Medical University
Locations (25):
- China (25):
  - Department of Anesthesiology, Beijing Obstetrics Gynecology Hospital, Beijing, Beijing Municipality
  - Departmet of Anesthesiology, Beijing Chao Yang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Department of Anesthesiology, China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Department of Anesthesioly,Peking University First Hospital, Beijing, Beijing Municipality
  - Department of Anesthesiology, Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Department of Anesthesiology, Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Department of Anesthesiology, Beijing Hangtian General Hospital, Beijing, Beijing Municipality
  - Department of Anesthesiology, Peking University Third Hospital, Beijing, Beijing Municipality
  - Department of Anesthesiology, Beijing Command General Hospital, Beijing, Beijing Municipality
  - Department of Anesthesiology, Beijing Hospital, Beijing, Beijing Municipality
  - Department of Anesthesiology, Beijing Tongren Hospital, Beijing, Beijing Municipality
  - Department of Anesthesiology, Fuzhou General Hospital, Fuzhou, Fujian
  - Department of Anesthesiology, Guangzhou first people ' s hospital, Guangzhou, Guangdong
  - Department of Anesthesiology, Nanfang Hospital, Guangzhou, Guangdong
  - Department of Anesthesiology, Wuhan Union Hospital, Wuhan, Hubei
  - Department of Anesthesiology, Xiangya Hospital of Central South University, Changsha, Hunan
  - Department of Anesthesiology, the First Hospital of Jilin University, Changchun, Jilin
  - Department of Anesthesiology, The First Hospital of China Medical University, Shenyang, Liaoning
  - Department of Anesthesiology, Shanghai Rui Jin Hospital, Shanghai, Shanghai Municipality
  - Department of Anesthesiology, Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Department of Anesthesiology, Shanghai Xinhua Hospital, Shanghai, Shanghai Municipality
  - Department of Anesthesiology, Second Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi’an, Shanxi
  - Department of Anesthesiology, Xijing Hospital, FMMU, Xi’an, Shanxi
  - Department of Anesthesiology, First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi’an, Shanxi
  - Department of Anesthesiology, Ningbo Lihuili Hospital, Ningbo, Zhejiang

REFERENCES:
- [Derived] Xu L, Wu AS, Yue Y. The incidence of intra-operative awareness during general anesthesia in China: a multi-center observational study. Acta Anaesthesiol Scand. 2009 Aug;53(7):873-82. doi: 10.1111/j.1399-6576.2009.02016.x. Epub 2009 Jun 3. PMID 19496761